CLINICAL TRIAL: NCT03420924
Title: Thermal Suit With Forced-air Warming in Breast Cancer Surgery: A Randomized Clinical Investigation
Brief Title: Thermal Suit With Forced-air Warming in Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R17137
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-02

CONDITIONS: Hypothermia, Accidental
Keywords: intraoperative hypothermia; thermal suit; forced-air warming
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermal suit (Experimental)
  Interventions: Device: Thermal suit
- Conventional hospital clothes (Active Comparator)
  Interventions: Device: Conventional hospital clothes

INTERVENTIONS:
Device: Thermal suit — Forced-air warming device will be connected to the trouser legs of the thermal suit.
  Arms: Thermal suit
Device: Conventional hospital clothes — The warming mattress and a forced-air warming blanket for the lower body will be used intraoperatively.
  Arms: Conventional hospital clothes

SUMMARY:
The aim of this clinical investigation is to prove that the thermal suit with forced-air warming is more effective to prevent inadvertent intraoperative hypothermia than conventional warming methods. The study group will have the thermal suit from arriving to the hospital until to the ward after surgery. In the operating theatre forced-air warming device will be connected to the trouser legs of the thermal suit and the device will be turned on during surgery. The control group will have normal hospital clothes. Intraoperative warming will be managed with the warming mattress and a forced-air warming blanket. The primary endpoint is core temperature after arriving to the post-anaesthesia care unit.

ELIGIBILITY:
Inclusion Criteria:

* primary breast cancer surgery
* unilateral resection or mastectomy with or without axillar lymphadenectomy
* body mass index 25-40

Exclusion Criteria:

* ASA > III
* decreased mental status
* inadequate Finnish language skills
* other than general anaesthesia

Ages: 20 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
Core temperature | 1 hour
  Core temperature after arriving to the post-anaesthesia care unit

CONTACTS AND LOCATIONS:
Overall Officials: Maija-Liisa Kalliomäki, Study Director — Tampere University Hospital
Locations (1):
- TAYS Hatanpää, Tampere, Finland